CLINICAL TRIAL: NCT03488108
Title: A Randomized Controlled Trial Comparing Platelet Rich Plasma (PRP) to Minoxidil Foam for Treatment of Androgenic Alopecia in Women
Brief Title: Platelet Rich Plasma Versus Minoxidil Foam for Treatment of Androgenic Alopecia in Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alison J. Bruce, Associate Professor of Dermatology, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-003335
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Alopecia
Keywords: growth factors, hair loss, females, regenerative therapy
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma first, then Minoxidil Foam (Experimental): Subjects will be randomized into the Platelet Rich Plasma group, treated for 12 weeks with a 2 month washout period in between treatments, then treated with Minoxidil Foam for 12 weeks.
  Interventions: Other: Platelet Rich Plasma; Drug: Minoxidil Foam
- Minoxidil Foam first, then Platelet Rich Plasma (Experimental): Subjects will be randomized into the Minoxidil Foam group, treated for 12 weeks with a 2 month washout period in between treatments, then treated with Platelet Rich Plasma.
  Interventions: Other: Platelet Rich Plasma; Drug: Minoxidil Foam

INTERVENTIONS:
Other: Platelet Rich Plasma — Autologous Platelet Rich Plasma (PRP) will be isolated from blood collected from each subject at each treatment time point. 100 cc of PRP will be injected with a 30-gauge needle over the affected part of the scalp, approximately 1/10 cc/injection site. Treatments will take place every 4 weeks for a total of 3 treatments over 12 weeks.
Drug: Minoxidil Foam — Minoxidil 5% topical foam will be applied once daily following manufacturer's instructions for a total of 12 weeks.
  Other Names: Rogaine

SUMMARY:
The primary objective of this proposal is to conduct a study that assesses the safety, feasibility and efficacy of using PRP to treat this type of hair loss.

DETAILED DESCRIPTION:
Androgenic alopecia (AGA) is a common, progressive hair loss disorder affecting both sexes with significant negative impact on social and psychological well-being. The frequency and severity increases with age, and up to 80% of men, and 50% of women are affected by AGA over the course of their lives. While men are more frequently affected, the psychological impact is likely to be high for women where the social impact of hair loss is often devastating. Current medical therapies specifically approved by the US FDA are limited to minoxidil (for men and women) and finasteride (for men only) (Varothai), but variable responses and the need for indefinite use often result in patient fatigue and suboptimal compliance. Recently, there has been interest in treatments orientated to more biologically regenerative therapies, and consequently there have been numerous studies that have demonstrated successful use for platelet rich plasma (PRP) in treating AGA. PRP contains concentrated platelet cells derived from autologous whole blood that are believed to activate a cascade of growth factors when injected into an area of poor hair growth that stimulates hair growth. In this proposal we will examine whether PRP therapy provides similar or better hair growing capacity in women compared to the conventional topical application minoxidil.

ELIGIBILITY:
Inclusion Criteria:

1. Only female patients are eligible
2. Patients must be 18 years of age or older
3. Patients must have Androgenic Alopecia Grade I-II by Ludwig Classification
4. Patients must have been on stable birth control if premenopausal.
5. Patients are able and willing to provide written informed consent after the nature of the study is fully explained

Exclusion Criteria:

1. Patients with clinically abnormal hematology, serum chemistry, or screening laboratory results as reviewed by the Principal Investigator
2. Patients who have undergone topical and systemic therapies for hair loss 3 months prior to the procedure
3. Patients who have used any cosmetic product meant to address hair loss 3 months prior to enrollment
4. Patients taking anti-rheumatic disease medication (including methotrexate or other anti-metabolites) within the 3 months prior to study entry.
5. Patients previously having undergone hair transplant surgery prior to study entry
6. Patients who are pregnant or currently breast-feeding children as Rogaine for Women is contra indicated for these women
7. Patients who have taken spironolactone in the 3 months prior to study participation
8. Patients with systemic, rheumatic or inflammatory disease or who are immunosuppressed
9. Patients with ongoing infectious disease, including HIV and hepatitis
10. Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer, or diabetes
11. Patients participating in a study of an experimental drug or medical device within 30 days of study entry
12. Patients with history of platelet disorders, bone marrow aplasia, sepsis, or cancer in the last 5 years.
13. Patients taking antiaggregating therapy
14. Patients on anticoagulant therapy
15. Patients with tendency to keloid formation
16. Patients with uncompensated diabetes
17. Patients with active skin disease or skin infection at intended treatment areas

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Bruce, M.B. Ch.B, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruce AJ, Pincelli TP, Heckman MG, Desmond CM, Arthurs JR, Diehl NN, Douglass EJ, Bruce CJ, Shapiro SA. A Randomized, Controlled Pilot Trial Comparing Platelet-Rich Plasma to Topical Minoxidil Foam for Treatment of Androgenic Alopecia in Women. Dermatol Surg. 2020 Jun;46(6):826-832. doi: 10.1097/DSS.0000000000002168. PMID 31574029
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet Rich Plasma First, Then Minoxidil Foam: Subjects who received PRP in either the first or last 12 weeks of the study
  Subjects will be randomized into the Platelet Rich Plasma group, treated for 12 weeks with a 2 month washout period in between treatments, then treated with Minoxidil Foam for 12 weeks.
  Platelet Rich Plasma: Autologous Platelet Rich Plasma (PRP) will be isolated from blood collected from each subject at each treatment time point. 100 cc of PRP will be injected with a 30-gauge needle over the affected part of the scalp, approximately 1/10 cc/injection site. Treatments will take place every 4 weeks for a total of 3 treatments over 12 weeks.
  Minoxidil Foam: Minoxidil 5% topical foam will be applied once daily following manufacturer's instructions for a total of 12 weeks.
- Minoxidil Foam First, Then Platelet Rich Plasma: Subjects who received Minoxidil either the first or last 12 weeks of the study
  Subjects will be randomized into the Minoxidil Foam group, treated for 12 weeks with a 2 month washout period in between treatments, then treated with Platelet Rich Plasma.
  Platelet Rich Plasma: Autologous Platelet Rich Plasma (PRP) will be isolated from blood collected from each subject at each treatment time point. 100 cc of PRP will be injected with a 30-gauge needle over the affected part of the scalp, approximately 1/10 cc/injection site. Treatments will take place every 4 weeks for a total of 3 treatments over 12 weeks.
  Minoxidil Foam: Minoxidil 5% topical foam will be applied once daily following manufacturer's instructions for a total of 12 weeks.
Period: First Intervention (12 Weeks)
Arm/Group | Platelet Rich Plasma First, Then Minoxidil Foam | Minoxidil Foam First, Then Platelet Rich Plasma
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (2 Months)
Arm/Group | Platelet Rich Plasma First, Then Minoxidil Foam | Minoxidil Foam First, Then Platelet Rich Plasma
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Platelet Rich Plasma First, Then Minoxidil Foam | Minoxidil Foam First, Then Platelet Rich Plasma
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phototrichogram Analysis, Vellus Hair Density, Quality of Life (QoL)
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma First, Then Minoxidil Foam | Minoxidil Foam First, Then Platelet Rich Plasma | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 51 [20 to 79] | 56 [20 to 79] | 56 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Hair Count
Description: Phototrichograms of all scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the total number of hairs per 0.65 cm2 was measured after both interventions, in each Arm/Group.
Time Frame: baseline, after 12 weeks of treatment
Population: One subject dropped out of the study after received PRP treatment only. This subject is included in results information regarding PRP only.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Platelet Rich Plasma: Subjects who received PRP in either the first or last 12 weeks of the study.
- Minoxidil Foam: Subjects who received Minoxidil either the first or last 12 weeks of the study.
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 18
percent change | 7.7 [-7.2 to 17.9] | 22.7 [-18.0 to 59.0]
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Minoxidil Foam; Test type: Superiority; p = .009, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Vellus Hair Density
Description: Phototrichograms of all scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the total number of vellus hairs per cm2 was measured after both interventions, in each Arm/Group.
Time Frame: baseline, after 12 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 18
percent change | 25.7 [-37.6 to 121.3] | 18.6 [-29.4 to 166.5]
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Minoxidil Foam; Test type: Superiority; p = .90, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Terminal Hair Density
Description: Phototrichograms of all scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the total number of Terminal hairs per cm2 was measured after both interventions, in each Arm/Group.
Time Frame: baseline, after 12 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 18
percent change | -0.7 [-49.5 to 27.6] | 12.8 [-19.4 to 119.4]
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Minoxidil Foam; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Cumulative Thickness
Description: Phototrichograms of all scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the total sum of thickness of each hair was measured after both interventions, in each Arm/Group.
Time Frame: baseline, after 12 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 18
percent change | -3.5 [-14.1 to 32.2] | 20.6 [-21.3 to 83.3]
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Minoxidil Foam; Test type: Superiority; p = .005, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Adverse Event of Swelling on Scalp
Description: Total number of participants experiencing swelling on scalp was measured after both interventions, in each Arm/Group.
Time Frame: after 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

6. Secondary Outcome: Adverse Event of Redness on Scalp
Description: Total number of participants experiencing Redness on Scalp was measured after both interventions, in each Arm/Group.
Time Frame: after 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during first treatment period, washout period, second treatment period and follow up period for a total of approximately 1 year.
Arm/Group | Platelet Rich Plasma | Minoxidil Foam
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 3/19 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (N=19) | Minoxidil Foam (N=18)
Pain (General disorders) | 2 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03488108/Prot_SAP_000.pdf